CLINICAL TRIAL: NCT05146336
Title: CytOSorb TreatMent Of Critically Ill PatientS Registry: International Registry on the Use of CytoSorb in the Critical Care Setting
Brief Title: CytOSorb TreatMent Of Critically Ill PatientS Registry
Acronym: COSMOS
Status: Recruiting | Type: Observational
Sponsor: CytoSorbents, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: O06
Record Dates: First submitted 2021-11-23; First posted 2021-12-06 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Septic Shock; Acute Respiratory Distress Syndrome; Trauma; Rhabdomyolysis; Cardiogenic Shock; Pancreatitis; Acute on Chronic Liver Failure; Acute Liver Failure; Burns; Chimeric Antigen Receptor T-Cell Therapy (CAR-T) Cytokine Release Syndrome (CRS); Extracorporeal Life Support; Postoperative Endocarditis; Hemophagocytic Lymphohistiocytoses; Liver Transplant; Complications; Infectious Disease; Postoperative Vasoplegic Syndrome; Drug Overdose; Sepsis
MeSH Terms: conditions — Shock, Septic; Respiratory Distress Syndrome; Wounds and Injuries; Rhabdomyolysis; Shock, Cardiogenic; Pancreatitis; Acute-On-Chronic Liver Failure; Liver Failure, Acute; Burns; Cytokine Release Syndrome; Lymphohistiocytosis, Hemophagocytic; Communicable Diseases; Vasoplegia; Drug Overdose; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: CytoSorb — Sorbent hemoperfusion system

SUMMARY:
Registry intended to provide a data repository and reporting infrastructure for the surveillance of CytoSorb device use in real-world critical care settings, and to serve as an objective, comprehensive, and scientifically-based resource to measure and improve the quality of patient care

ELIGIBILITY:
Inclusion Criteria:

1. Planned OR actual CytoSorb® 300 mL device utilization
2. Informed consent for prospective registry participation

Exclusion Criteria:

1. Use of the CytoSorb® 300 mL device for antithrombotic removal only
2. Intraoperative use of CytoSorb® 300 mL device during cardiac surgery only
3. The occurrence of a complication or other medically justified circumstance that arises after written informed consent has been obtained from the patient and before or during the planned therapy and as a result of which the use of CytoSorb® 300 mL Adsorber is contraindicated or no longer appropriate.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Critically ill patients receiving CytoSorb therapy
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2022-06-22 (Actual); Primary Completion 2032-06 (Estimated); Study Completion 2032-09 (Estimated)

PRIMARY OUTCOMES:
ICU mortality | Through ICU discharge or date of death, whichever comes first [on average 7 days]
In-hospital mortality | Through hospital discharge or date of death, whichever comes first [on average 14 days]

CONTACTS AND LOCATIONS:
Overall Officials: Ricard Ferrer Roca, MD, Principal Investigator — Hospital Vall d'Hebron
Locations (28):
- Austria (2):
  - Klinikum Klagenfurt am Wörthersee, Klagenfurt
  - Medizinische Universität Wien, Vienna
- Germany (18):
  - Universitätsklinikum Aachen, Aachen
  - Herz- und Diabeteszentrum Nordrhein-Westfalen, Bad Oeynhausen
  - Berufsgenossenschaftliches Universitätsklinikum Bergmannsheil Bochum, Bochum
  - Katholisches Klinikum Bochum, St. Josef-Hospital, Bochum
  - Universitätsklinikum Essen, Medizinische Intensivtherapie, Essen
  - Universitätsklinikum Essen, Nephrologie, Essen
  - Universitätsklinikum Essen, Thorax- und Kardiovaskuläre Chirurgie, Essen
  - Universitätsmedizin Göttingen, Allgemein-, Viszeral- und Kinderchirurgie, Göttingen
  - Universitätsmedizin Göttingen, Herzzentrum Göttingen, Göttingen
  - Klinikum Herford, Herford
  - Universitätsklinikum Jena, Jena
  - Klinikum Kassel, Kassel
  - Universitätsklinikum Marburg, Marburg
  - Kliniken Maria Hilf, Mönchengladbach
  - Deutsches Herzzentrum München, München
  - LMU Klinikum München, München
  - Klinikum Oldenburg, Oldenburg
  - Helios Dr. Horst Schmidt Kliniken Wiesbaden, Wiesbaden
- Italy (2):
  - Ospedale Pediatrico Bambino Gesù, Roma
  - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
- Poland (2):
  - SP ZOZ Szpital Uniwersytecki w Krakowie, Krakow
  - Uniwersyteckim Spitalem Klinicznym im. Jana Mikulicza - Radeckiego we Wrocławiu, Wroclaw
- Portugal (2):
  - Unidade Local de Saúde de Coimbra E.P.E, Coimbra
  - ULS São José, Hospital Curry Cabral, Lisbon
- Spain (2):
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona
  - Hospital Juan Ramón Jimenez, Huelva

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ferrer R, Thielmann M, Kribben A, Unglaube M, Tyczynski B, Kreutz J, Baumann A, Guenther U, Henzler D, Kirschning T, El-Essawi A, Gunther T, Bellgardt M, Bottari G, Aucella F, Hidalgo J, Teboul JL, Tomescu D, Klaus T, Fan W, Scheier J, Deliargyris EN, Taccone FS. The international, prospective CytOSorbⓇ treatMent Of critically ill patientS (COSMOS) registry: Interim results from the first 150 patients. J Intensive Med. 2025 Jun 27;5(4):392-399. doi: 10.1016/j.jointm.2025.05.001. eCollection 2025 Oct. PMID 41180104
- [Derived] Taccone FS, Brunkhorst FM, Bottari G, Hidalgo J, Kribben A, Teboul JL, Tomescu D, Klaus T, Scheier J, Deliargyris E, Ferrer R. The COSMOS Registry of CytoSorb Hemoadsorption Therapy in Critically Ill Patients: Protocol for an International, Prospective Registry. JMIR Res Protoc. 2024 Nov 5;13:e55880. doi: 10.2196/55880. PMID 39500494